CLINICAL TRIAL: NCT02366637
Title: A Randomized, Double-blind, Placebo-controlled 2-way Crossover Study To Evaluate The Efficacy, Safety And Tolerability Of Pf-03715455 Administered Twice Daily By Inhalation For 4 Weeks In Subjects With Moderate To Severe Chronic Obstructive Pulmonary Disease (Copd)
Brief Title: An Evaluation Of PF-03715455 In Moderate To Severe Chronic Obstructive Pulmonary Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated on 7 April 2015 for business reasons. No safety and/or efficacy concerns contributed to the termination of the study
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: A9111004; INHALED p38i COPD; 2014-002340-40 (EudraCT Number)
Record Dates: First submitted 2014-09-02; First posted 2015-02-19 (Estimated); Results first posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Sputum
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — N-(1-(3-chloro-4-hydroxyphenyl)-3-(1,1-dimethylethyl)-1H-pyrazol-5-yl)-N'-((2-((3-(2-((2-hydroxyethyl)thio)phenyl)-1,2,4-triazolo(4,3-a)pyridin-6-yl)thio)phenyl)methyl)-urea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Double blind placebo for PF-03715455
  Interventions: Drug: Placebo
- PF-03715455 (Experimental)
  Interventions: Drug: PF-03715455

INTERVENTIONS:
Drug: Placebo — Orally inhaled placebo twice a day (BID) for 4 weeks
  Arms: Placebo
Drug: PF-03715455 — 680 micrograms BID, Orally inhaled PF-03715455 for 4 weeks
  Arms: PF-03715455

SUMMARY:
This study proposes to evaluate the safety and efficacy of PF-03715455 in subjects with moderate to severe Chronic Obstructive Pulmonary Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of non-childbearing potential and male subjects between the ages of 40 and 80 years, inclusive
* Subjects with a diagnosis, for at least 6 months, of moderate to severe COPD and who meet the criteria for Stage II-III disease
* Subjects must have a smoking history of at least 10 pack-years

Exclusion Criteria:

* Current evidence or history within the previous 6 months of any clinically significant disease (other than COPD) or abnormality in the opinion of the Investigator that would put the subject at risk or which would compromise the quality of the study data
* A COPD exacerbation requiring treatment with oral steroids or hospitalization for the treatment of COPD within 3 months of Screening

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United Kingdom (5):
  - Medicines Evaluation Unit Ltd, Wythenshawe, Manchester
  - Nottingham University Hospital NHS Trust, Nottingham, Nottinghamshire
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Heart of England NHS Foundation Trust, Birmingham
  - Respiratory Medicine, Bradford Institute of Health Research, Bradford

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9111004&StudyName=An%20Evaluation%20Of%20PF-03715455%20In%20Moderate%20To%20Severe%20Chronic%20Obstructive%20Pulmonary%20Disease

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomly assigned in a 1:1 ratio to receive either PF-03715455 680 micrograms (mcg) twice daily for 4 weeks or matching placebo in Period 1. Participants who were randomized to PF-03715455 during Period 1 then received placebo for 4 weeks during Period 2 after a 28 to 49-day washout period, and vice versa.
Groups:
- PF-03715455 680 mcg Twice Daily: PF-03715455 680 mcg dry powder capsule was administered by oral inhalation twice daily via a Miat mondose inhaler device for 4 weeks in each treatment period. Dosing in each treatment period was separated by a washout period of 28 to 49 days.
- Placebo: Matching placebo was administered by oral inhalation twice daily via a Miat mondose inhaler device for 4 weeks in each treatment period. Dosing in each treatment period was separated by a washout period of 28 to 49 days.
Period: First Intervention Period
Arm/Group | PF-03715455 680 mcg Twice Daily | Placebo
Started | 7 | 6
Completed | 1 | 1
Not Completed | 6 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Study Terminated by Sponsor | 6 | 4
Period: Washout Period 28 to 49 Days
Arm/Group | PF-03715455 680 mcg Twice Daily | Placebo
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0
Period: Second Intervention Period
Arm/Group | PF-03715455 680 mcg Twice Daily | Placebo
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Study Terminated by Sponsor | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants who received at least 1 dose of study drug (PF-03715455 or placebo).
Arm/Group | All Participants
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) at Week 4
Description: FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. Trough FEV1 was obtained from spirometry, performed before study treatment administration.
Time Frame: Baseline (Day 1), Day 29 (Week 4)
Population: The modified intent-to-treat (mITT) analysis set included all randomized participants who received at least 1 dose of study drug; n=number of participants analyzed in respective arms for category.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | PF-03715455 680 mcg Twice Daily | Placebo
Number analyzed (Participants) | 8 | 7
liters
  Baseline (n=8,7) | 1.368 (0.3534) | 1.456 (0.5209)
  Change at Week 4 (n=6,6) | -0.047 (0.0983) | 0.080 (0.2310)

2. Secondary Outcome: Change From Baseline in Sputum Cell Counts Over 4 Weeks
Description: Sputum cell counts included total neutrophils counts and differential (percent [%]), total cell count, total macrophage count and differential (%). Change over 4 weeks was to be presented.
Time Frame: Baseline, Week 1 to Week 4
Population: It was not meaningful to summarize sputum cell counts as there were too few participants in the sputum sub-study and, of those, too few adequate sputum specimens to be meaningfully summarized.
Arm/Group | PF-03715455 680 mcg Twice Daily | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in Trough FEV1 and Forced Vital Capacity (FVC) at Weeks 1, 3, and 4
Description: FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. FVC is the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. FEV1 Baseline and Change at Week 4 are already reported under Primary Outcome Measure 1.
Time Frame: Baseline, Day 7 (Week 1), Day 21 (Week 3), Day 29 (Week 4)
Population: The mITT analysis set included all randomized participants who received at least 1 dose of study drug; n=number of participants analyzed in respective arms for category.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | PF-03715455 680 mcg Twice Daily | Placebo
Number analyzed (Participants) | 8 | 7
liters
  FEV1: Change at Week 1 (n=8,7) | -0.065 (0.1231) | -0.001 (0.2559)
  FEV1: Change at Week 3 (n=8,7) | -0.039 (0.2194) | -0.026 (0.1033)
  FVC: Baseline (n=8,7) | 2.535 (0.8639) | 3.263 (1.2571)
  FVC: Change at Week 1 (n=8,7) | -0.019 (0.1336) | 0.090 (0.1630)
  FVC: Change at Week 3 (n=8,7) | 0.049 (0.2100) | -0.079 (0.1893)
  FVC: Change at Week 4 (n=6,6) | 0.091 (0.1661) | 0.233 (0.3014)

4. Secondary Outcome: Change From Baseline in Trough FEV1 and Forced Vital Capacity (FVC) Over 4 Weeks
Description: FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. FVC is the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Change over 4 weeks is presented.
Time Frame: Baseline, Week 1 to Week 4
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | PF-03715455 680 mcg Twice Daily | Placebo
Number analyzed (Participants) | 8 | 7
liters
  FEV1: Change Over 4 Weeks (n=6,6) | -0.047 (0.0983) | 0.080 (0.2310)
  FVC: Change Over 4 Weeks (n=6,6) | 0.091 (0.1661) | 0.233 (0.3014)

5. Secondary Outcome: Maximum Observed Plasma Concentrations (Cmax) of PF-03715455
Time Frame: Pre-dose on Day 7 and Day 21; post-dose on Day 7 (10 minutes and 1 hour post-dose) and Day 29
Population: As pharmacokinetics (PK) was not a primary objective of the study, only sparse PK sampling was performed to allow for a population PK analysis. As the study was prematurely terminated, there were too few subjects to perform this analysis. Therefore, the PK was not analyzed.
Arm/Group | PF-03715455 680 mcg Twice Daily
Number analyzed (Participants) | 0

6. Secondary Outcome: Trough Plasma Concentration (Ctrough) of PF-03715455
Description: Ctrough is the concentration prior to study drug administration.
Time Frame: Pre-dose on Day 7 and Day 21; post-dose on Day 7 (10 minutes and 1 hour post-dose) and Day 29
Population: As PK was not a primary objective of the study, only sparse PK sampling was performed to allow for a population PK analysis. As the study was prematurely terminated, there were too few subjects to perform this analysis. Therefore, the PK was not analyzed.
Arm/Group | PF-03715455 680 mcg Twice Daily
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Day 29 that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to Day 29 (Week 4)
Population: The mITT analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | PF-03715455 680 mcg Twice Daily | Placebo
Number analyzed (Participants) | 8 | 7
participants
  AEs | 3 | 4
  SAEs | 0 | 0

8. Other Pre Specified Outcome: Number of Participants With Clinically Significant Treatment Emergent Electrocardiogram (ECG) Findings
Description: Clinically significant ECG findings include: PR interval >=300 milliseconds (msec) or >=25% increase when baseline is >200 msec and >=50% increase when baseline is less than or equal to 200 msec; QRS interval >=200 msec or >=25/50% increase from baseline; QT interval >=500 msec; corrected QT interval using Fridericia's formula (QTcF) >=450 msec or >=30 msec increase.
Time Frame: Baseline up to Day 29 (Week 4)
Population: The mITT analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | PF-03715455 680 mcg Twice Daily | Placebo
Number analyzed (Participants) | 8 | 7
participants
  PR Interval >=300 msec | 0 | 0
  QRS Complex >=200 msec | 0 | 0
  QT Interval >=500 msec | 0 | 0
  QTcF Interval 450-<480 msec | 0 | 0
  QTcF Interval 480-<500 msec | 0 | 0
  QTcF Interval >=500 msec | 0 | 0
  PR Interval >=25/50% Increase From Baseline | 0 | 0
  QRS Complex >=25/50% Increase From Baseline | 0 | 0
  QTcF Interval 30-<60 msec Increase From Baseline | 0 | 0
  QTcF Interval >=60 msec Increase From Baseline | 0 | 0

9. Other Pre Specified Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure
Description: Systolic blood pressure (SBP) and diastolic pressure (DBP) were evaluated in the supine position.
Time Frame: Baseline, Day 7 (Week 1), Day 21 (Week 3), Day 29 (Week 4), Day 49 (follow-up)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | PF-03715455 680 mcg Twice Daily | Placebo
Number analyzed (Participants) | 8 | 7
millimeters of mercury (mmHg)
  SBP: Baseline (n=8,7) | 130.0 (19.16) | 122.7 (13.92)
  SBP: Change at Week 1 (n=7,6) | -7.4 (13.24) | 1.3 (3.01)
  SBP: Change at Week 3 (n=5,5) | -3.4 (12.03) | -0.6 (9.02)
  SBP: Change at Week 4 (n=8,7) | -2.0 (15.34) | 8.1 (7.06)
  SBP: Change at Follow-Up (n=7,6) | 1.4 (13.49) | 4.7 (11.24)
  DBP: Baseline (n=8,7) | 69.9 (9.72) | 65.1 (9.01)
  DBP: Change at Week 1 (n=7,6) | 0.6 (6.95) | 8.7 (8.69)
  DBP: Change at Week 3 (n=5,5) | 2.4 (7.09) | 4.4 (5.13)
  DBP: Change at Week 4 (n=8,7) | 2.1 (3.91) | 2.4 (8.46)
  DBP: Change at Follow-Up (n=7,6) | 5.4 (6.63) | 2.8 (5.04)

10. Other Pre Specified Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate was evaluated in the supine position.
Time Frame: Baseline, Day 7 (Week 1), Day 21 (Week 3), Day 29 (Week 4), Day 49 (follow-up)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | PF-03715455 680 mcg Twice Daily | Placebo
Number analyzed (Participants) | 8 | 7
beats per minute (bpm)
  Baseline (n=8,7) | 66.5 (11.82) | 64.3 (9.71)
  Change at Week 1 (n=7,6) | 3.6 (7.41) | 3.5 (3.56)
  Change at Week 3 (n=5,5) | -1.6 (3.36) | 0.0 (3.16)
  Change at Week 4 (n=8,7) | 1.3 (2.96) | 1.3 (6.24)
  Change at Follow-Up (n=7,6) | 2.0 (4.76) | 1.0 (3.35)

11. Other Pre Specified Outcome: Number of Participants With Laboratory Abnormalities
Description: The following laboratory parameters were analyzed: hematology (hemoglobin, hematocrit, red blood cell [RBC] count, RBC morphology, platelet count, white blood cell [WBC] count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); blood chemistry (blood urea nitrogen [BUN], creatinine, glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase [AST], alanine aminotransferase [ALT], total bilirubin, direct and indirect bilirubin, gamma-glutamyl transpeptidase [GGT], alkaline phosphatase, uric acid, albumin, total protein, high sensitivity C-reactive protein [CRP]); urinalysis (specific gravity, pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, microscopy [only if urine dipstick was positive for blood or protein]).
Time Frame: Baseline up to Week 4
Population: The mITT analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | PF-03715455 680 mcg Twice Daily | Placebo
Number analyzed (Participants) | 8 | 7
participants | 6 | 4

ADVERSE EVENTS:
Time Frame: Baseline up to follow-up period (Day 49)
Arm/Group | PF-03715455 680 mcg Twice Daily | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 3/8 | 4/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | PF-03715455 680 mcg Twice Daily (N=8) | Placebo (N=7)
Palpitations (Cardiac disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1/3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
As this study was prematurely terminated by the sponsor for business reasons, no formal safety or efficacy conclusions can be drawn due to insufficient participant numbers. In addition, PK analysis was not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.